CLINICAL TRIAL: NCT02440594
Title: The PACE/PACENET Behavioral Health Laboratory Project: Evaluation of a Clinical Management Program Among Older Adults Newly Prescribed Medication for Behavioral Health Issues
Brief Title: The PACE/PACENET Behavioral Health Laboratory Project
Acronym: SUSTAINII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Magellan Health Services (Other)
Responsible Party: Principal Investigator, David Oslin, Professor of Psychiatry, Department of Psychiatry, Perelman School of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 807774
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-09

CONDITIONS: Depression
Keywords: Primary Care; Depression; Elderly
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Enhanced Care High-Symptom AD/AX (Experimental): Patients newly prescribed an antidepressant or anxiolytic who report significant baseline symptoms receive Enhanced BHL Program Services, which include the: 1) Standard Clinical Monitoring Module - evidence-based care consisting of up to 4 brief (5-10 minutes), structured assessments following the Core/baseline assessment. Interviews are conducted over the telephone by the Health Technician/BHP and take place during the initial 12 weeks of pharmaceutical treatment (e.g., 2, 6, 9, and 12 weeks), and monitor adherence, side effects, and treatment response. A progress report is provided to the prescribing clinician after each interview to help in treatment planning and to alert the clinician of special issues, and 2) Enhanced Care Management Module - Care Management services with a BHP.
  Interventions: Behavioral: Enhanced BHL Program Services
- Standard Care High-Symptom AD/AX (Active Comparator): Patients newly prescribed an antidepressant or anxiolytic who report significant baseline symptoms receive Standard BHL Program Services, which include the Standard Clinical Monitoring Module - evidence-based care consisting of up to 4 brief (5-10 minutes), structured assessments following the Core/baseline assessment. Interviews are conducted over the telephone by the Health Technician/BHP and take place during the initial 12 weeks of pharmaceutical treatment (e.g., 2, 6, 9, and 12 weeks), and monitor adherence, side effects, and treatment response. A progress report is provided to the prescribing clinician after each interview to help in treatment planning and to alert the clinician of special issues.
  Interventions: Behavioral: Standard BHL Program Services
- Enhanced Monitoring Low-Symptom AD/AX/AP (Experimental): Patients newly prescribed an antidepressant, anxiolytic, or antipsychotic who report low baseline symptoms receive Enhanced BHL Program Services, which for this group include the: 1) Standard Clinical Monitoring Module - evidence-based care consisting of up to 4 brief (5-10 minutes), structured assessments following the Core/baseline assessment. Interviews are conducted over the telephone by the Health Technician/BHP and take place during the initial 12 weeks of pharmaceutical treatment (e.g., 2, 6, 9, and 12 weeks), and monitor adherence, side effects, and treatment response. A progress report is provided to the prescribing clinician after each interview to help in treatment planning and to alert the clinician of special issues, and 2) Enhanced Monitoring via a one-time BHP follow-up call with the enrollee after 6 weeks to discuss continuing versus discontinuing the medication.
  Interventions: Behavioral: Enhanced BHL Program Services
- Standard Monitoring Low-Symptom AD/AX/AP (Active Comparator): Patients newly prescribed an antidepressant, anxiolytic, or antipsychotic who report low baseline symptoms receive Standard BHL Program Services, which include the Standard Clinical Monitoring Module - evidence-based care consisting of up to 4 brief (5-10 minutes), structured assessments following the Core/baseline assessment. Interviews are conducted over the telephone by the Health Technician/BHP and take place during the initial 12 weeks of pharmaceutical treatment (e.g., 2, 6, 9, and 12 weeks), and monitor adherence, side effects, and treatment response. A progress report is provided to the prescribing clinician after each interview to help in treatment planning and to alert the clinician of special issues.
  Interventions: Behavioral: Standard BHL Program Services
- Enhanced Care High-Symptom AP (Experimental): Patients newly prescribed an antipsychotic who report significant baseline symptoms receive Enhanced BHL Program Services, which include the: 1) Standard Clinical Monitoring Module - evidence-based care consisting of up to 4 brief (5-10 minutes), structured assessments following the Core/baseline assessment. Interviews are conducted over the telephone by the Health Technician/BHP and take place during the initial 12 weeks of pharmaceutical treatment (e.g., 2, 6, 9, and 12 weeks), and monitor adherence, side effects, and treatment response. A progress report is provided to the prescribing clinician after each interview to help in treatment planning and to alert the clinician of special issues, and 2) Enhanced Care Management Module - Care Management services with a BHP.
  Interventions: Behavioral: Enhanced BHL Program Services
- Standard Care High-Symptom AP (Active Comparator): Patients newly prescribed an antipsychotic who report significant baseline symptoms receive Standard BHL Program Services, which include the Standard Clinical Monitoring Module - evidence-based care consisting of up to 4 brief (5-10 minutes), structured assessments following the Core/baseline assessment. Interviews are conducted over the telephone by the Health Technician/BHP and take place during the initial 12 weeks of pharmaceutical treatment (e.g., 2, 6, 9, and 12 weeks), and monitor adherence, side effects, and treatment response. A progress report is provided to the prescribing clinician after each interview to help in treatment planning and to alert the clinician of special issues.
  Interventions: Behavioral: Standard BHL Program Services
- Caregiver TEP Intervention (Experimental): Caregivers of patients newly prescribed an antidepressant, anxiolytic, or antipsychotic who cannot participate due to cognitive impairment and meet criteria for dementia receive Enhanced BHL Program Services which include: 1) a baseline clinical assessment of caregiver and care recipient factors (e.g., level of disability, burden, safety concerns) and contact information for local community services, and 2) the Telehealth Education Program (TEP) - BHPs provide manual and workbook-guided psychoeducation, support, and skills training.
  Interventions: Behavioral: Enhanced BHL Program Services
- Caregiver Control (Active Comparator): Caregivers of patients newly prescribed an antidepressant, anxiolytic, or antipsychotic who cannot participate due to cognitive impairment and meet criteria for dementia receive Standard BHL Program Services, which include a baseline clinical assessment of caregiver and care recipient factors (e.g., level of disability, burden, safety concerns) and contact information for local community services
  Interventions: Behavioral: Standard BHL Program Services

INTERVENTIONS:
Behavioral: Enhanced BHL Program Services — Patients or their caregivers will work with a BHP to provided additional support and education beyond the services received in the Standard BHL Program.
  Arms: Caregiver TEP Intervention; Enhanced Care High-Symptom AD/AX; Enhanced Care High-Symptom AP; Enhanced Monitoring Low-Symptom AD/AX/AP
Behavioral: Standard BHL Program Services — Patients or their caregivers receive a baseline clinical assessment as well as monitoring of symptoms and referral to community resources.
  Arms: Caregiver Control; Standard Care High-Symptom AD/AX; Standard Care High-Symptom AP; Standard Monitoring Low-Symptom AD/AX/AP

SUMMARY:
The purpose of the current project is to conduct a program evaluation that examines the impact of the The SUpporting Seniors Receiving Treatment And INtervention (SUSTAIN) program - a telephone-based clinical service designed to help identify and manage behavioral health issues among enrollees in the Commonwealth of Pennsylvania Department of Aging's Pharmaceutical Assistance Contract for the Elderly and the PACE Needs Enhancement Tier Program (PACE/PACENET) - on enrollee outcomes and to evaluate the feasibility and impact of an enhancement to the current clinical program.

DETAILED DESCRIPTION:
Despite advances in the assessment and treatment of behavioral health disorders among older adults, such disorders remain inadequately diagnosed and managed in later life. This is troubling in light of the fact that behavioral health issues often serve as the catalyst for a variety of negative psychosocial and physical health outcomes in later life, including changes in social network functioning, physical disability and morbidity, loss of independence, and institutionalization. Factors such as limited provider resources for conducting frequent monitoring, variability in patient preferences and symptom severity, patients' lack of treatment acceptance and engagement, low medication adherence, formal and informal social support and aid, and logistic issues (e.g., transportation, finances, etc.) all work in concert to influence patient identification and disease management. Yet, these factors are difficult to address when managing conditions using traditional mental health (MH) care delivery models that rely primarily on referrals to specialty care and/or face-to-face contact.

Recognizing that traditional MH care delivery models and treatment strategies do not address both practice- and patient-level logistical issues that are particularly relevant in behavioral health care, where frequent clinical visits for monitoring and therapeutic contact are key components in the successful treatment of patients, the investigators have adopted a strategy of delivering disease management by way of telephone assessments. The Behavioral Health Laboratory (BHL) is a flexible and dynamic telephone-based clinical service designed to help identify and manage behavioral health issues. The principles of the program include: MH as a key component to overall physical health; the need to make early MH screening, assessment, and referral to services a part of common practice; the value in utilizing technology in accessing and delivering MH care; and the importance of research- and evidence-based practice.

An untoward outcome of the efforts to improve rates of treatment is the increased and sometimes inappropriate use of psychotropic medication. Among the general population, the use of psychotropic medication and rates of psychotropic polypharmacy continue to rise, with increased use of medication for both anxiety and depression in both primary care and specialty care. The rates of use have raised concerns regarding inappropriate prescribing among the elderly.

Results from the investigators' initial program of care management services for PACE/PACENET cardholders support the above concerns related to psychotropic medication prescription in the elderly and also raise additional questions about off-label or inappropriate prescribing. The program results indicate that the PACE/PACENET population is mostly female with a mean age of 78.1 years (SD 7.0), and an SF-12 Physical Component Score of 41.6. The average Patient Health Questionnaire-9 (PHQ-9) score for those on antidepressants (AD) was 6.1 (5.4), with no statistically significant difference between medication groups (F(2.436)=2.14, p=0.12); just 9 (6.3%) of those receiving anxiolytics (AX) met criteria for an anxiety disorder, which was not significantly different than other medication classes (x2(2)=1.77, p=0.41). Overall, 208 (47.4%) participants in the sample did not meet criteria for any mental health disorder, including 80 (55.9%) of those receiving anxiolytics.

Thus, the purpose of the current project is to evaluate the impact of the PACE/PACENET BHL clinical programs on older Pennsylvanians and to evaluate the feasibility and impact of enhancements to the current clinical program. The clinical contract for services targets PACE/PACENET beneficiaries who have been newly prescribed an antidepressant, antipsychotic (AP), and/or anxiolytic, and, where appropriate, their caregivers. In order to obtain a representative sample of PACE/PACENET enrollees, the PACE/PACENET program uses a stratified sampling method for the identification and referral of eligible beneficiaries to the PACE/PACENET BHL Clinical Program. Stratification is conducted with respect to two variables--county and medication type, with individuals randomly selected from each strata. Current clinical participants are not being sampled or contacted specifically for research purposes. The research portion of this project relates only to the evaluation of those enrolled in the clinical program and to the delivery and evaluation of the enhancements to the current program. Moreover, while the program provides services to a variety of patients with varying types and levels of symptoms, our primary objectives are specific to patients prescribed an antidepressant or anxiolytic who show significant baseline symptomatology. Nonetheless, we describe all program participants below.

The PACE/PACENET BHL Research Participants:

1. Enhanced BHL Program Participants:

   Upon completion of the initial PACE/PACENET BHL Program interview, the investigators will randomly select a subset of up to 2400 enrollees for the Enhanced BHL Program and invite the enrollees to participate in the Enhanced Program. If the enrollee is not able to complete the full initial BHL interview due to cognitive impairment (either as identified by cognitive screening or caregiver report), the caregiver may be invited to participate in the caregiver component of the Enhanced BHL Program, the Telehealth Education Program (TEP) Module.
2. BHL Program Evaluations: Participants recruited for the evaluation component of the BHL Programs (Standard and Enhanced) will fall into the following categories:

   1. Evaluation of BHL Clinical Data: In order to examine factors such as participant clinical and sociodemographic characteristics, process of care, prescription refills, and use of services, the investigators will ask enrollees for permission to use the clinical data collected during the BHL interviews. To accomplish this component of the evaluation, the investigators will orally consent all individuals who at least begin a Core interview to allow use of the clinical data for research purposes. Participants do not need to consent to use of the clinical data as a prerequisite to participating in the clinical program. The clinical data will include their prescription data supplied by the PACE/PACENET program.
   2. 3/6 Month Outcome Evaluation: In order to examine long-term outcomes, participants who complete an initial clinical interview will be offered participation in an outcome evaluation at 3 and 6 months.

Subject Recruitment and Screening:

1. BHL Clinical Data Evaluation: Following completion of the initial PACE/PACENET BHL clinical assessment (i.e., "Core assessment"), all enrollees will be asked for permission to use the clinical data collected during the BHL interviews.
2. Enhanced Program Recruitment: Following completion of the initial PACE/PACENET BHL clinical assessment, a subset of enrollees will be asked to participate in the Enhanced BHL Program. Randomization to the Enhanced Program will occur within strata as determined by index medication type and Core interview assessment outcome (i.e., clinically significant depression and/or anxiety symptoms, no clinically significant symptoms, cognitive impairment). After obtaining informed consent, a separate simple randomization protocol will be followed within each substratum of enrollees. For each substratum every other participant will be offered participation in the Enhanced BHL Program.
3. 3/6 Month Outcome Evaluation Recruitment: Following completion of the initial PACE/PACENET clinical assessments and agreement to participation in the Enhanced Program or our Standard Clinical Program, enrollees or the caregivers will be asked to participate in an evaluation of the BHL program at 3 and 6 months from the initial PACE/PACENET BHL clinical interview.

Study Procedures:

The Enhanced BHL Program:

1. The Enhanced BHL Program: Upon completion of the Core interview, a subset of enrollees will be randomly selected to participate in the Enhanced BHL Program (i.e., Enhanced Monitoring Module or Enhanced Care Management Module). For enrollees who do not report clinically significant mental health symptoms the Enhanced Program consists of the Standard Monitoring Module enhanced with a discussion of continuing versus discontinuing the medication. The Behavioral Health Provider (BHP) will follow-up with the enrollee after 6 weeks to discuss continuing versus discontinuing the medication. For enrollees who report clinically significant depression, anxiety, and/or pain symptoms the Enhanced Program consists of Care Management. The model incorporates the use of a BHP who has expertise in mental health assessment and is well versed in the delivery of algorithm-based management strategies for disorders such as depression and anxiety. The role of the BHP is to facilitate treatment and provide informal psychosocial therapy, using motivational interviewing techniques, in a manner that is consistent with the Agency for Health Care Policy and Research (AHCPR) guidelines. The BHP monitors and encourages patient acceptance and adherence to treatment recommendations through support, education, and motivational engagement. The BHP initiates care management when enrollees are not responding to the initial treatment or as clinically needed based on the initial Core interview and needs assessment. The BHP also uses problem solving therapy to assist patients. In cases where caregivers participate due to the enrollees' cognitive impairment, they will be asked to participate in the Telehealth Education Program (TEP). The TEP is a manual-driven psychosocial support and skills training program for caregivers of individuals with moderate to severe cognitive impairment. The frequency and number of contacts for each individual will vary; individuals typically engage in 1-2 contacts per month for several months. Written updates are provided to the prescribing clinician, as clinically indicated.
2. 3/6 Month Outcome Evaluation: In order to evaluate individual-level outcomes and rates of clinical improvement at 3 and 6 months, the investigators will attempt to collect follow-up data from all enrollees/caregivers who have completed the initial PACE/PACENET BHL Clinical Program assessment. Using data extracted from the enrollee follow-up assessments, the investigators will examine psychological, behavioral, and cognitive symptoms, physical disability, health care utilization, and access to community resources. Using data extracted from caregiver follow-up assessments, the investigators will be able to evaluate care recipients' behavioral, psychological, and cognitive symptoms and level of physical functioning, in addition to caregiver burden and safety concerns.

ELIGIBILITY:
Inclusion Criteria:

1. To be eligible for the Enhanced BHL Program, the only inclusion criterion is to have participated in an initial telephone assessment as part of the current PACE/PACENET BHL Clinical Program.
2. Similarly, to be eligible for the BHL Program Evaluations (i.e., BHL Clinical Data Evaluation, 3/6 Month Outcome Evaluation), the inclusion criterion is to have participated in an initial telephone assessment as part of the current PACE/PACENET BHL Clinical Program.
3. Enrollment in the current PACE/PACENET BHL Clinical Program. Though not part of the research program, the current program targets older, community-dwelling adults (i.e., 65 years and older) enrolled in the PACE/PACENET programs, who have filled at least one new prescription for an antidepressant, antipsychotic, and/or anxiolytic medication. The BHL program does require the basic ability to communicate by telephone; either the enrollee or an identified caregiver must meet this criterion for participation in the BHL Clinical Program.

Exclusion Criteria:

Exclusion criteria for participation in the Enhanced BHL Program and the 3/6 Month Outcome Evaluation are:

1. having severe cognitive impairment (BOMC score 14 or greater) in the absence of a caregiver, and/or
2. endorsement of psychosis or mania during the initial clinical interview, and/or
3. a PHQ score of 25 or greater, and/or
4. positive drug abuse screen, and/or
5. alcohol dependence.

Enrollees endorsing any of above mentioned exclusions will be offered assistance with referral to community specialty-care resources as part of the PACE/PACENET BHL Clinical Program.

Exclusion criteria for caregiver participation in the TEP component of Enhanced Care is lack of report of cognitive impairment when only the Caregiver interview was completed.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2432 (Actual)
Dates: Start 2010-08; Primary Completion 2014-11 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W Oslin, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Department of Psychiatry (Addictions/Geriatric), University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Oslin DW, Ross J, Sayers S, Murphy J, Kane V, Katz IR. Screening, assessment, and management of depression in VA primary care clinics. The Behavioral Health Laboratory. J Gen Intern Med. 2006 Jan;21(1):46-50. doi: 10.1111/j.1525-1497.2005.0267.x. PMID 16423122
- [Background] Maust DT, Mavandadi S, Eakin A, Streim JE, Difillipo S, Snedden T, Oslin DW. Telephone-based behavioral health assessment for older adults starting a new psychiatric medication. Am J Geriatr Psychiatry. 2011 Oct;19(10):851-8. doi: 10.1097/JGP.0b013e318202c1dc. PMID 21946801
- [Result] Maust DT, Mavandadi S, Benson A, Streim JE, Difilippo S, Snedden T, Weber AL, Oslin DW. Telephone-based care management for older adults initiated on psychotropic medication. Int J Geriatr Psychiatry. 2013 Apr;28(4):410-6. doi: 10.1002/gps.3839. Epub 2012 Jun 7. PMID 22678956
- [Result] Maust DT, Chen SH, Benson A, Mavandadi S, Streim JE, DiFilippo S, Snedden TM, Oslin DW. Older adults recently started on psychotropic medication: where are the symptoms? Int J Geriatr Psychiatry. 2015 Jun;30(6):580-6. doi: 10.1002/gps.4187. Epub 2014 Aug 12. PMID 25116369
- [Result] Mavandadi S, Benson A, DiFilippo S, Streim JE, Oslin D. A Telephone-Based Program to Provide Symptom Monitoring Alone vs Symptom Monitoring Plus Care Management for Late-Life Depression and Anxiety: A Randomized Clinical Trial. JAMA Psychiatry. 2015 Dec;72(12):1211-8. doi: 10.1001/jamapsychiatry.2015.2157. PMID 26558530

RESULTS

PARTICIPANT FLOW:
Recruitment Details: To conduct the program evaluation, clinical record data were extracted for patients (newly prescribed an antidepressant (AD), anxiolytic (AX), or antipsychotic (AP)) and caregivers enrolled in the SUSTAIN (SUpporting Seniors Receiving Treatment And INtervention) program between 8/5/10 and 5/15/14 who completed a baseline clinical interview.
Groups:
- Enhanced Care High-Symptom AD/AX: Patients newly prescribed an antidepressant or anxiolytic who report significant baseline symptoms receive Enhanced BHL Program Services, which include the: 1) Standard Clinical Monitoring Module - evidence based care consisting of up to 4 brief (5-10 minutes), structured assessments following the Core/baseline assessment. Interviews are conducted over the telephone by the Health Technician/BHP and take place during the initial 12 weeks of pharmaceutical treatment (e.g., 2, 6, 9, and 12 weeks), and monitor adherence, side effects, and treatment response. A progress report is provided to the prescribing clinician after each interview to help in treatment planning and to alert the clinician of special issues, and 2) Enhanced Care Management Module - Care Management services with a BHP.
Period: Overall Study
Arm/Group | Enhanced Care High-Symptom AD/AX | Standard Care High-Symptom AD/AX | Enhanced Monitoring Low-Symptom AD/AX/AP | Standard Monitoring Low-Symptom AD/AX/AP | Enhanced Care High-Symptom AP | Standard Care High-Symptom AP | Caregiver TEP Intervention | Caregiver Control
Started | 509 | 509 | 436 | 429 | 55 | 54 | 150 | 290
Completed (Completed numbers reflect number completing 2 or more follow-ups assessments) | 377 | 401 | 319 | 340 | 46 | 47 | 113 | 234
Not Completed | 132 | 108 | 117 | 89 | 9 | 7 | 37 | 56
Not completed — Lost to Follow-up | 34 | 33 | 54 | 47 | 5 | 4 | 28 | 48
Not completed — Cognitive Impairment/Communication Issue | 14 | 6 | 4 | 4 | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 81 | 67 | 59 | 38 | 2 | 2 | 7 | 7
Not completed — Administratively w/drawn | 3 | 2 | 0 | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Includes SUSTAIN program participants who completed a baseline clinical assessment and enrolled in program services.
Groups:
- Enhanced Monitoring Low-Symptom AD/AX/AP: Patients newly prescribed an antidepressant, anxiolytic, or antipsychotic who report low baseline symptoms receive Enhanced BHL Program Services, which for this group include the: 1) Standard Clinical Monitoring Module - evidence-based care consisting of up to 4 brief (5-10 minutes), structured assessments following the Core/baseline assessment. Interviews are conducted over the telephone by the Health Technician/ BHP and take place during the initial 12 weeks of pharmaceutical treatment (e.g., 2, 6, 9, and 12 weeks), and monitor adherence, side effects, and treatment response. A progress report is provided to the prescribing clinician after each interview to help in treatment planning and to alert the clinician of special issues, and 2) Enhanced Monitoring via a one-time BHP follow-up call with the enrollee after 6 weeks to discuss continuing versus discontinuing the medication.
- Total: Total of all reporting groups
Arm/Group | Enhanced Care High-Symptom AD/AX | Standard Care High-Symptom AD/AX | Enhanced Monitoring Low-Symptom AD/AX/AP | Standard Monitoring Low-Symptom AD/AX/AP | Enhanced Care High-Symptom AP | Standard Care High-Symptom AP | Caregiver TEP Intervention | Caregiver Control | Total
Number analyzed (Participants) | 509 | 509 | 436 | 429 | 55 | 54 | 150 | 290 | 2432
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.7 (6.8) | 77.4 (6.7) | 78.1 (6.6) | 78.1 (6.5) | 76.6 (6.7) | 74.7 (6.9) | 63.3 (11.9) | 64.3 (12.0) | 77.6 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 440 | 407 | 364 | 352 | 41 | 43 | 114 | 208 | 1969
  Male | 69 | 102 | 72 | 77 | 14 | 11 | 36 | 82 | 463
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 472 | 467 | 405 | 390 | 54 | 53 | 132 | 265 | 2238
  Other | 37 | 42 | 31 | 39 | 1 | 1 | 18 | 25 | 194
Region of Enrollment [Number; unit: participants]
  United States | 509 | 509 | 436 | 429 | 55 | 54 | 150 | 290 | 2432

OUTCOME MEASURES:

1. Primary Outcome: Medical Outcomes Survey Short Form (SF12) Mental Component Subscale (MCS) Score
Description: A measure of overall mental health functioning as measured by the Medical Outcomes Survey Short Form (SF12) MCS subscale. Possible range = 0-100; higher scores mean better overall health functioning.
Time Frame: Baseline and 3 and 6 month follow-up
Population: SUSTAIN participants who were prescribed an AD or AX (per pharmacy records) and endorsed high baseline MH symptoms during the initial clinical interview. This was not a primary outcome measure for those patients assigned to the other 4 groups; data were extracted from clinical records only for patients assigned to the two designated arms.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Care High-Symptom AD/AX | Standard Care High-Symptom AD/AX
Number analyzed (Participants) | 509 | 509
score on a scale
  Baseline | 47.52 (11.15) | 48.94 (10.14)
  3 month follow-up: number analyzed (Participants) | 352 | 328
  3 month follow-up | 51.03 (10.34) | 51.11 (9.97)
  6 month follow-up: number analyzed (Participants) | 352 | 330
  6 month follow-up | 51.92 (10.07) | 50.35 (10.58)

2. Primary Outcome: Zarit Burden Interview (ZBI)
Description: Brief, 4-item version of the Zarit Burden Interview; Possible range = 0-16; higher scores denote greater perceived caregiving burden. This measure was only collected of caregivers who participated in SUSTAIN program services.
Time Frame: Baseline and 3 and 6 month follow-up
Population: Caregivers who completed a baseline clinical interview and agreed to SUSTAIN caregiver services.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver TEP Intervention | Caregiver Control
Number analyzed (Participants) | 150 | 290
score on a scale
  Baseline | 6.54 (4.00) | 5.37 (4.34)
  3 month follow-up: number analyzed (Participants) | 94 | 205
  3 month follow-up | 5.57 (4.03) | 5.36 (4.36)
  6 month follow-up: number analyzed (Participants) | 92 | 180
  6 month follow-up | 5.37 (3.52) | 5.36 (4.22)

3. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: A 9-item measure of depressive symptom severity in past 2 weeks. Possible range = 0-27; higher scores indicate higher depressive symptom severity.
Time Frame: Baseline and 3 and 6 month follow-up
Population: Analyses run for SUSTAIN program participants who were prescribed, 1) an AD or AX and endorsed high baseline MH symptoms during the initial clinical interview and, 2) an AP and endorsed high baseline MH symptoms. Due to their low baseline symptom severity, these outcome data were only collected/extracted at baseline for the low symptom groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Care High-Symptom AD/AX | Standard Care High-Symptom AD/AX | Enhanced Care High-Symptom AP | Standard Care High-Symptom AP | Enhanced Monitoring Low-Symptom AD/AX/AP | Standard Monitoring Low-Symptom AD/AX/AP
Number analyzed (Participants) | 509 | 509 | 55 | 54 | 436 | 429
score on a scale
  Baseline | 8.83 (4.56) | 8.64 (4.27) | 10.07 (5.14) | 10.33 (5.26) | 1.78 (1.44) | 1.79 (1.42)
  3 month follow-up: number analyzed (Participants) | 356 | 332 | 42 | 37 | 0 | 0
  3 month follow-up | 5.70 (4.48) | 6.04 (4.72) | 7.45 (4.97) | 6.57 (6.28) |  |
  6 month follow-up: number analyzed (Participants) | 356 | 336 | 38 | 40 | 0 | 0
  6 month follow-up | 5.68 (4.57) | 6.82 (4.91) | 7.55 (4.12) | 8.38 (6.44) |  |

4. Secondary Outcome: Generalized Anxiety Disorder - 7 (GAD-7)
Description: A 7-item measure of anxiety symptom severity over the past 2 weeks. Possible range = 0 - 21; higher scores indicated greater anxiety symptom severity
Time Frame: Baseline and 3 and 6 month follow-up
Population: SUSTAIN participants prescribed an antidepressant or anxiolytic and endorsed high baseline MH symptoms during the initial clinical interview. Due to their different symptom profiles and index medications, these outcome data were only collected/extracted at baseline for the low symptom and AP groups, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Care High-Symptom AD/AX | Standard Care High-Symptom AD/AX | Enhanced Care High-Symptom AP | Standard Care High-Symptom AP | Enhanced Monitoring Low-Symptom AD/AX/AP | Standard Monitoring Low-Symptom AD/AX/AP
Number analyzed (Participants) | 509 | 509 | 55 | 54 | 436 | 429
units on a scale
  Baseline | 4.75 (4.41) | 4.48 (4.21) | 5.85 (5.17) | 6.41 (5.29) | 0.88 (1.20) | 0.79 (1.07)
  3 month follow-up: number analyzed (Participants) | 356 | 330 | 0 | 0 | 0 | 0
  3 month follow-up | 3.09 (3.72) | 3.42 (3.82) |  |  |  |
  6 month follow-up: number analyzed (Participants) | 355 | 336 | 0 | 0 | 0 | 0
  6 month follow-up | 2.79 (3.61) | 3.90 (4.34) |  |  |  |

5. Secondary Outcome: Number of Participants With Moderately Severe to Severe Depression (Per Patient Health Questionnaire-9 (PHQ-9))
Description: Number of participants with moderately severe to severe depression at Baseline, 3 and 6 months; Depression diagnosis (i.e., moderately severe - severe depression vs. no - minimal depression or minor - moderate depression) based on a 9-item measure of depressive symptom severity in past 2 weeks.
Time Frame: Baseline and 3 and 6 month follow-up
Population: Numbers represent number of participants in each low symptom arm who met criteria for moderately severe - severe depression at 3 and 6 months. Due to their different symptom profiles, these outcome data were only collected/extracted at baseline for the high symptom groups.
Measure: Number; unit: participants
Arm/Group | Enhanced Monitoring Low-Symptom AD/AX/AP | Standard Monitoring Low-Symptom AD/AX/AP | Enhanced Care High-Symptom AD/AX | Standard Care High-Symptom AD/AX | Enhanced Care High-Symptom AP | Standard Care High-Symptom AP
Number analyzed (Participants) | 436 | 429 | 509 | 509 | 55 | 54
participants
  Baseline | 0 | 0 | 62 | 55 | 11 | 15
  3 month follow-up: number analyzed (Participants) | 285 | 249 | 0 | 0 | 0 | 0
  3 month follow-up | 5 | 6 |  |  |  |
  6 month follow-up: number analyzed (Participants) | 284 | 242 | 0 | 0 | 0 | 0
  6 month follow-up | 6 | 5 |  |  |  |

ADVERSE EVENTS:
Time Frame: 6 months
Description: The research assessment for program evaluation purposes was only done at 3 and 6 months post-randomization; adverse events were not recorded as part of the program evaluation and only death would have been noted at the time of the 3 or 6 month assessments.
Groups:
- Standard Monitoring Low-Symptom AD/AX/AP: Patients newly prescribed an antidepressant, anxiolytic, or antipsychotic who report low baseline symptoms receive Standard BHL Program Services, which include the Standard Clinical Monitoring Module - evidence based care consisting of up to 4 brief (5-10 minutes), structured assessments following the Core/baseline assessment. Interviews are conducted over the telephone by the Health Technician/BHP and take place during the initial 12 weeks of pharmaceutical treatment (e.g., 2, 6, 9, and 12 weeks), and monitor adherence, side effects, and treatment response. A progress report is provided to the prescribing clinician after each interview to help in treatment planning and to alert the clinician of special issues.
Arm/Group | Enhanced Care High-Symptom AD/AX | Standard Care High-Symptom AD/AX | Enhanced Monitoring Low-Symptom AD/AX/AP | Standard Monitoring Low-Symptom AD/AX/AP | Enhanced Care High-Symptom AP | Standard Care High-Symptom AP | Caregiver TEP Intervention | Caregiver Control
All-Cause Mortality (participants affected / at risk) | 12/509 | 10/509 | 2/436 | 6/429 | 3/55 | 1/54 | 0/150 | 1/290
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No